CLINICAL TRIAL: NCT04083040
Title: Impact of Tilt Angle on Conduction Defects During Transcatheter Aortic Valve Implantation (TAVI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Moubasher, DR, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tilt angle during TAVI
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: TAVI
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVI patients (Other): Patient undergone TAVI
  Interventions: Procedure: transcatheter aortic valve implantation

INTERVENTIONS:
Procedure: transcatheter aortic valve implantation — 1. Tilt angle.
  2. Depth of implantation of the valve.
  3. Type of the valve.(Medtronic core valve self expandable valve ,Edwards sapient balloon expandable valve

SUMMARY:
Investigate the predictors of conduction abnormalities after TAVI, and in particular the predictive role of the tilt-angle during implantation.

DETAILED DESCRIPTION:
The method of transcatheter aortic valve implantation (TAVI) which was introduced in 2002 by Alain Cribier et al. has offered new prospects for patients with severe aortic stenosis and multiple comorbidities, for whom surgical procedures are associated with exceedingly high operative risk (1,2).

The randomized multicenter PARTNER trial (Placement of Aortic Transcatheter valve Trial) proved that TAVI is an alternative for surgical aortic valve replacement (SAVR) for high-risk patients.TAVI is characterized by similar mortality and results in terms of reducing the symptoms of stenosis (3).

Current recommendations by the European Society of Cardiology in the Guidelines on the management of valvular heart disease (4) are that TAVI should be carried out in patients with a life expectancy >1 year, who deemed inoperable or high-risk by a cardiac surgeon and who are likely to gain improvement in quality of life. (5).

One of the complications based on the consensus of experts (the Valve Academic Research Consortium-2 (VARC-2 criteria)) is Conduction defect (6).

The mechanical interaction of the prosthesis stent frame with the conduction system and left bundle branch may lead to a high degree of or complete AV block and to left bundle branch block (LBBB) after TAVI.(7)

The pathophysiology of new conduction abnormalities has not yet been elucidated. A number of studies indicate that both patient and procedure related factors such as septal wall thickness, non-coronary cusp thickness, pre-existing RBBB, depth of valve implantation within the LVOT, post implant prosthesis expansion, and the type of prosthesis play a role , LVOT/ annulus ratio, LVOT/Prosethesis diameter..(8)(9)(10)(11)(12)

ELIGIBILITY:
Inclusion Criteria:

* 1- Intermediate or high risk patient for surgical aortic valve replacement ,EuroSCORE >15% or an STS score >10%. (13)

  2- Transfermoral approach.

  2- Contraindications for open chest surgery, such as(14) :

Expected high perioperative risk due to comorbidities not adequately reflected by scores :

1. Squelae of chest radiation.
2. Severe chest deformation or scoliosis.
3. Previous cardiac surgery

Exclusion Criteria:

* A- Clinical conditions.

  1. Active endocarditis,
  2. Myocardial infarction within 14 days
  3. Cardiogenic shock
  4. Life expectancy of less than 1 year.
  5. Patients with previously implanted Permenant Pacemakers.

B- Anatomical conditions:

1. short distance between coronary ostia and aortic valve annulus.
2. Size of aortic annulus out of range for TAVI(range from 18mm - 27mm)(14).
3. Elevated risk of coronary ostium obstruction (asymmetric valve calcification, short distance between annulus and coronary ostium, small aortic sinuses).
4. Plaques with mobile thrombi in the ascending aorta, or arch. For transfemoral/subclavian approach: inadequate vascular access (vessel size, calcification, tortuosity).
5. left Ventricular Thrombus.

C-Severe primary associated disease of other valves or significant coronary artery disease with major contribution to the patient's symptoms that can be treated only by surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
TILT ANGLE | 1 year
  Investigate the predictors of conduction abnormalities after TAVI, and in particular the predictive role of the tilt-angle during implantation.